CLINICAL TRIAL: NCT01173419
Title: A Multi-Center, Randomized, Controlled Study to Evaluate the Efficacy and Safety of Subjects Comparing the NeverTouch Versus the RF ClosureFAST Methods of Treatment of the Great Saphenous Vein
Brief Title: Comparison Study for Safety and Efficacy of Two Devices for the Treatment of the Great Saphenous Vein
Acronym: RECoN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision to reevaluate clinical needs.
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PV-201
Record Dates: First submitted 2010-07-28; First posted 2010-08-02 (Estimated); Last update posted 2012-07-13 (Estimated); Status verified 2012-07

CONDITIONS: Varicose Veins; Venous Insufficiency
Keywords: Great Saphenous Vein
MeSH Terms: conditions — Varicose Veins; Venous Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VenaCure EVLT NeverTouch (Active Comparator)
  Interventions: Device: VenaCure EVLT NeverTouch
- RF ClosureFAST (Active Comparator)
  Interventions: Device: VNUS RF ClosureFAST

INTERVENTIONS:
Device: VNUS RF ClosureFAST — VNUS® RF ClosureFAST is a minimally invasive varicose vein treatment procedure that uses radiofrequency energy (electricity) to heat, collapse and seal off the targeted blood vessels.
  Other Names: Closure
  Arms: RF ClosureFAST
Device: VenaCure EVLT NeverTouch — Endovenous Laser Treatment (EVLT) uses laser energy, which is a highly concentrated beam of light to treat varicose veins.
  Other Names: VenaCure; EVLT; NeverTouch
  Arms: VenaCure EVLT NeverTouch

SUMMARY:
This is a multi center, randomized, comparison study using two already cleared methods of treatment of the great saphenous vein (GSV). The hypothesis to be tested is that the use of the Venacure EVLT NeverTouch procedure is no worse than the RF ClosureFAST procedure for treatment of the GSV. Evaluation of post operative pain and bruising, quality of life assessments, adverse event assessments, confirmation of long term GSV closure, use of medications are criteria that will be evaluated during the course of this study.

DETAILED DESCRIPTION:
Some form of venous insufficiency affects up to 25% of men and 40% of women in the United States. While most persons seek treatment because varicose veins are unsightly, most will also experience symptoms such as aching pain, night cramps, leg fatigue, leg heaviness or leg restlessness. If left untreated, nearly 50% of patients with significant superficial venous insufficiency will experience chronic venous insufficiency characterized by lower extremity swelling, eczema, pigmentation, hemorrhage and ulceration.

This is a multicenter, prospective, randomized study in subjects with symptomatic venous insufficiency of the great saphenous vein. Subjects evaluated for participation will be those who, prior to the first visit, have elected to receive invasive treatment for the GSV insufficiency and have already received conservative treatment (i.e. use of compression hose).

Subjects will be randomized to receive one of two methods of treatment. VenaCure EVLT NeverTouch method of treatment or the RF ClosureFAST method of treatment.

Follow up visits will take place at 2, 7, 14 and 30 days post treatment where questionnaires (SF-36, CIVI Q2, Visual Analogue Scale), evaluation of GSV closure via duplex ultrasound (7 day and 30 day only), evaluation of ecchymosis, physician (or their designee) evaluation of venous disease (CEAP assessment and VCSS assessment), assessments of adverse events and review of concomitant medications (use of analgesics and other medications)will take place. These same evaluations with the exception of the use of the Visual Analogue Scale and the Ecchymosis evaluation will also take place at the 6 month and 12 month follow up visit timepoints.

ELIGIBILITY:
Inclusion Criteria:

* male or female,
* 18 to 80 years of age,
* have documented symptomatic GSV disease defined by any of the following:
* C2 disease
* C3 disease
* C4A, C4B disease
* C5 disease
* C6 disease
* have not been previously treated for GSV,
* have multilevel venous reflux in the great saphenous vein greater than 0.5 seconds after distal compression/ release in the standing position,
* have palpable dorsalis pedis/ anterior tibial pulse or ABI >0.9 (unless calcified pressures) at screening,
* are able to comply with the protocol requirements,
* are able to comprehend and willing to sign an Informed Consent Form (ICF).

Exclusion Criteria:

* has had a previous venous intervention on the same leg as planned current treatment,
* are in a known hypercoagulable state,
* have deep vein thrombosis or a history of deep vein thrombosis,
* have thrombus within the last three months in the vein segment to be treated,
* have an aneurysmal section in the vein segment to be treated (aneurysm is defined as 2 times greater than the adjacent vein),
* are not able to ambulate,
* have non staged adjunctive procedures such as sclerotherapy and/ or ambulatory phlebectomy. May elect to stage the procedure from the initial script, and not treat before the 30 day follow up visit is completed.
* are, in the opinion of the investigator, unable to comply with the schedule and protocol evaluations,
* are currently pregnant or breast feeding,
* have a known malignancy other than skin cancer,
* current use of anticoagulant medication,
* have any condition which in the opinion of the investigator could compromise subject safety or adherence to the protocol,
* has had treatment with any investigational agent within 30 days of visit 1.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of post operative adverse events/ effects between the two treatment groups. | Evaluated on the day of treatment (post treatment), 2, 7, 14, and 30 days and 6 and 12 months post treatment follow up visits.

SECONDARY OUTCOMES:
Evaluation of GSV closure and incidence of DVT via duplex ultrasound between the two treatment groups. | Evaluated at 7 and 30 days post treatment and 6 and 12 months post treatment follow up visits.
Presence and intensity of post operative pain between the two treatment groups. | Evaluated at 2, 7, 14 and 30 days and 6 and 12 months post treatment follow up visits.
  The VAS scale for pain will be used through the 30 day follow up time period. The questionnaires for quality of life will be used for each of the visits including the 6 and 12 month follow up visits.
Presence and intensity of post operative ecchymosis between the two treatment groups. | Evaluated 2, 7, 14 and 30 days post treatment follow up visits.
  A blinded healthcare professional (selected by the PI at each site) will evaluate the subject at the designated timepoints.
Use of Analgesics within the 30 days post treatment between the two treatment groups. | Reviewed at 2, 7, 14 and 30 days post treatment follow up visits.
Evaluation of subject quality of life between the two treatment groups. | Completed at 2, 7, 14 and 30 days and 6 and 12 months post treatment follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: David Gillespie, MD, Principal Investigator — University of Rochester
Locations (6):
- United States (6):
  - UC Davis Interventional and Vascular Radiology, Sacramento, California
  - Batey Cardiovascular and Vein Center, Bradenton, Florida
  - Midwest Institute for Minimally Invasive Therapies (MIMIT), Melrose Park, Illinois
  - Novi Vein Center, Novi, Michigan
  - NYU Langone Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York